CLINICAL TRIAL: NCT07287072
Title: Pain Reprocessing Therapy for Chronic Primary Pain Caused by a Likely Nociplastic Pain Mechanism in Primary Care: The PRIME-PRT Trial
Brief Title: Pain Reprocessing Therapy for Chronic Primary Pain
Acronym: PRIME-PRT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Responsible Party: Principal Investigator, Silje Endresen Reme, Professor and psychologist, Oslo University Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 884238
Record Dates: First submitted 2025-12-02; First posted 2025-12-17 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Nociplastic Pain; Chronic Primary Pain
Keywords: chronic primary pain; Nociplastic pain; Pain Reprocessing Therapy
MeSH Terms: conditions — Nociplastic Pain; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Single Case Experimental Design (SCED). In a SCED study, the unit of analysis is the individual rather than the group, and the patient serves as their own control. Participants will be randomized to different starting periods for the intervention (Phase B) as soon as they are included in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRT (Experimental): Pain Reprocessing Therapy
  Interventions: Behavioral: Pain Reprocessing Therapy

INTERVENTIONS:
Behavioral: Pain Reprocessing Therapy — Pain Reprocessing Therapy (PRT) has shown promising results for patients with chronic primary back pain with a nociplastic pain-mechanism. PRT consists of two components. The first is an educational component (E) conducted by a physician. The purpose of the educational component is to reorient the patient's understanding of pain in accordance with the theories of nociplastic pain (false alarm based on negative expectations). The second part consists of a set of specific therapeutic techniques (T) that can be performed by a physician, psychologist, or other trained healthcare personnel. The techniques are easy to learn and have a training framework of 50 hours over a period of 3 months. They are based, among other things, on interoceptive exposure techniques, where the main point is to confront internal sensory experiences that have been interpreted as threatening (and ultimately lead to pain), with a new assurance that they do not signal danger ("false alarm").

SUMMARY:
Approximately 30% of adult Norwegians experience chronic pain, with its prevalence rising across demographics, including children and adolescents Chronic pain contributes to significant personal suffering and substantial societal costs. Traditional treatments - physical, pharmacological, and surgical - as well as psychological interventions, such as cognitive and acceptance-based therapies, demonstrate only minor to modest effects.

To address the challenge of rising demand alongside limited treatment options, university hospitals must consistently evaluate and adopt new, potentially effective therapies to meet their societal mission. Pain Reprocessing Therapy (PRT) is one such innovative treatment that has recently demonstrated promising results for a subset of chronic pain patients in a U.S. primary care setting.

In this study, the investigators want to assess the effectiveness of PRT on various outcomes in patients with primary chronic pain that has a likely nociplastic pain mechanism, within a Norwegian primary care population.

The insights from this study will be important for any prospective implementation of PRT to align with one of the guiding principles of the Norwegian healthcare system: the Best Effective Level of Care (BEON principle). The BEON principle supports the delivery of high-quality, cost-effective healthcare services and is founded on the notion of seamless integration across different levels of care. When competence or resources at the primary healthcare level are insufficient, more patients tend to be referred to higher, specialized, and inherently more costly levels of care, such as secondary and tertiary care. Therefore, if the study can demonstrate that PRT is effective within a Norwegian primary care population, the hypothesize is that its implementation could strengthen both primary and tertiary care in alignment with the BEON principle.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70
* On sick leave, or at risk of sick leave
* Pain intensity corresponding to 3 (or more) on the NRS from the PROMIS-29.
* Readiness to change, corresponding to the action stage from the readiness to change model, where they are ready to participate in their own change process

Exclusion Criteria:

* Structural causes for their pain (rheumatoid arthritis, cancer, etc.),
* Severe psychiatric conditions (ongoing or previous psychotic disorders, suicidality, or severe depression/anxiety/bipolar disorder)
* Illegal substance abuse, or known dependence on benzodiazepines or opioids
* Ongoing litigation or compensation process related to the pain condition
* Ongoing and severe psychosocial stressors (e.g. recent divorce etc.)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Average pain rating in the past 7 days on a numerical rating scale from 0-10 from Patient-Reported Outcomes Measurement Information System - 29 items (PROMIS-29) | 5-week post-treatment assessment (5 weeks after first PRT session; 1 week after final PRT session)
  Pain intensity average last week assessed through one item. The scale ranges from 0 (no pain) to 10 (worst imaginable pain)

SECONDARY OUTCOMES:
Physical function measured through PROMIS-29 | 5-week post-treatment assessment (5 weeks after first PRT session; 1 week after final PRT session) and at 1 year follow-up
  Patient-Reported Outcome Measurement Information System (PROMIS-29) average score post-treatment on the domain Physical function. Scores range from 4-20, with higher scores indicating better function
Individual goals assessed through Goal Attainment Scaling (GAS) | 5-week post-treatment assessment (5 weeks after first PRT session; 1 week after final PRT session) and at 1 year follow-up
  Individual goals as defined by the patient. For instance: "Running up a hill" or "playing basketball" (Ref to GAS: Ruble et al., 2012).
Work participation at 1-year follow-up | Assessed through self-report at 5 weeks follow-up and 1 year follow-up
  Increased work participation since baseline (y/n)
Patient Global Impression of Change | 5-week post-treatment assessment (5 weeks after first PRT session; 1 week after final PRT session)
  Patients' global impression of change in symptoms, function and quality of life (Hurst, 2004). The scale ranges from 1 (no change) to 7 (a great deal better and considerable improvement)

OTHER OUTCOMES:
Perceived injustice | Baseline, 5 weeks and 1 year follow-up
  Perceived injustice measured by Injustice Experience Questionnaire. The total score ranges from 0-48, with higher score indicating more perceived injustice.
Pain catastrophizing | Measured at 5 weeks post-treatment and at 1 year follow-up.
  Pain Catastrophizing Scale measured at 5 weeks post-treatment and at 1 year follow-up. The total score ranges from 0-52, where a higher score indicates more catastrophizing.
Fear of movement or re-injury | Measured 5 weeks post-treatment and at 1 year follow-up.
  Tampa Scale of Kinesiophobia (TSK-11). Scores range from 11 to 44, with higher score indicating more severe fear of movement.

CONTACTS AND LOCATIONS:
Locations (1):
- Ullevål sykehus, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
The investigators pan to share de-identified individual participant data with collaborating research groups in Sweden and the Netherlands. Access will be restricted to qualified researchers who submit an application and obtain approval from the relevant ethics committee and data protection authority. There is also a plan to share the study protocol, statistical analysis plan, and analysis code.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: From end of assessment (July 31st) and until December 31st 2027).
Access Criteria: Access will be restricted to qualified researchers who submit an application and obtain approval from the relevant ethics committee and data protection authority.

REFERENCES:
- [Background] Ashar YK, Gordon A, Schubiner H, Uipi C, Knight K, Anderson Z, Carlisle J, Polisky L, Geuter S, Flood TF, Kragel PA, Dimidjian S, Lumley MA, Wager TD. Effect of Pain Reprocessing Therapy vs Placebo and Usual Care for Patients With Chronic Back Pain: A Randomized Clinical Trial. JAMA Psychiatry. 2022 Jan 1;79(1):13-23. doi: 10.1001/jamapsychiatry.2021.2669. PMID 34586357